CLINICAL TRIAL: NCT02536157
Title: A Randomised Controlled Trial Investigating the Effectiveness of Two Splinting Methods in the Non-operative Management of Volar Plate Injuries at the Proximal Interphalangeal Joint
Brief Title: Volar Plate Injury: A Comparison of Two Splinting Methods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Health Service, United Kingdom (Other Government)
Collaborators: University of Bradford (Other)
Responsible Party: Principal Investigator, Claire Paxman, Senior Physiotherapist, National Health Service, United Kingdom
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 12020625
Record Dates: First submitted 2015-08-21; First posted 2015-08-31 (Estimated); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Volar Plate Injury of the Proximal Interphalangeal Joint
Keywords: Volar plate; Splint; Proximal interphalangeal joint; Palmar plate; Hyperextension injury

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dorsal block splint (Active Comparator): Thermoplastic splint in 20 degrees flexion applied to the dorsum of the PIPJ.
  Interventions: Device: Thermoplastic splinting
- Volar gutter splint (Experimental): Thermoplastic splint in 0 degrees flexion applied to the volar surface of the finger.
  Interventions: Device: Thermoplastic splinting

INTERVENTIONS:
Device: Thermoplastic splinting

SUMMARY:
Which splinting method produces the best outcomes (in range of movement, pain and function) in the non-operative treatment of stable volar plate injuries in adults?

The volar plate is a ligament located at the middle knuckle (proximal interphalangeal joint - PIPJ) of the finger. It is commonly injured through hyperextension, for example a ball hitting the fingertip. Current treatment in the Hand Therapy Unit involves splinting the injured joint dorsally (on the back of the finger) into 20⁰ flexion (bent) using thermoplastic material. However, there is a potential risk of developing permanent stiffness of the PIPJ into straightening, once the volar plate ligament heals. To reduce this risk, the study aims to investigate if using a volar (on the front of the finger) gutter splint in 0⁰ flexion (straight), which still prevents hyperextension, achieves better outcomes. There is no existing high-quality evidence comparing these two methods.

This is a randomised controlled trial. For the purposes of this study, the current treatment of a 20° dorsal block splint will act as the control group. The intervention group will be the volar gutter splint group. A convenience sample will be used and all patients (over 16 years old) presenting to the Mid Yorkshire Hospitals NHS Trust's Hand Therapy Unit will be invited to participate in the study, with consideration to inclusion/exclusion criteria. Participants will be randomised into one of two groups through the use of a random number generator. The outcomes assessed will be range of movement, pain and function. These will be measured at initial assessment, four and twelve weeks. These are all average normal time intervals that patients are seen. Each splint is worn for four weeks and participants will receive standardised advice, exercises and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. All stable volar plate injuries.
2. Aged 16 and older.
3. Male and female.
4. Acute presentation within 2 weeks of injury.
5. All ethnic groups speaking English.

Exclusion Criteria:

1. Vulnerable patient groups or those lacking capacity.
2. Previous injury or pathology involving the same digit.
3. Surgical intervention
4. Unstable proximal interphalangeal joint.
5. Concomitant tendon or additional bony injury outside the traditional Eaton classification types of volar plate injury.
6. The DASH outcome measure is available and validated in 27 languages. However, those who do not speak/understand English well will unfortunately be excluded. This is an educational project and therefore there is no funding to use a translator service.
7. Volar plate injuries are just as common in children and teenagers as adults. But under 16s will be excluded from this study as the DASH questionnaire has only been assumed valid in adults. There is no research investigating its use in younger age-groups.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Range of movement measured with a Jamar finger goniometer. | One week
  Range of movement measured with a Jamar finger goniometer.
Range of movement measured with a Jamar finger goniometer. | Four weeks
  Range of movement measured with a Jamar finger goniometer.
Range of movement measured with a Jamar finger goniometer. | Twelve weeks
  Range of movement measured with a Jamar finger goniometer.

SECONDARY OUTCOMES:
Pain measured using a 100mm visual analogue scale. | One, four and twelve weeks
  Measured using a 100mm visual analogue scale.
Function of the upper limb measured using the DASH questionnaire. | One, four and twelve weeks
  Disabilities of the Shoulder, Arm and Hand Questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Hand Therapy Unit, Mid Yorkshire Hospitals NHS Trust, Pinderfields General Hospital, Aberford Road,, Wakefield, West Yorkshire, United Kingdom